CLINICAL TRIAL: NCT06695650
Title: Investigating the Effect of Mandala Coloring Activity on Test Anxiety: A Randomized Controlled Trial
Brief Title: The Effect of Mandala Coloring Activity on Test Anxiety
Acronym: Mandala
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nursemin ÜNAL (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Sponsor-Investigator, Nursemin ÜNAL, Associate Professor, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/11
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Educational Problems; Anxiety; Test Anxiety; Mental Health
Keywords: Test anxiety; Nursing education; Mandala coloring; Randomized Controlled Trial
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single: The outcome assessor did not know which group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Group (Experimental): Students in the intervention group will be provided with mandala templates and coloring materials. They will be asked to color for 15 minutes twice a week over a two-month period. Email reminders will be sent to the students about the coloring sessions, and they will submit their completed mandalas to the researchers every Friday.
  "Demographic Characteristics Form" and a pre-test using the "Test Anxiety Inventory." Thirty minutes before the exam, the "Test Anxiety Inventory" will be applied as a post-test.
  Interventions: Other: Mandala Coloring
- Control Group (No Intervention): Non intervention. "Demographic Characteristics Form" and a pre-test using the "Test Anxiety Inventory." Thirty minutes before the exam, the "Test Anxiety Inventory" will be applied as a post-test.

INTERVENTIONS:
Other: Mandala Coloring — Students in the intervention group will be provided with mandala templates and coloring materials. They will be asked to color for 15 minutes twice a week over a two-month period
  Arms: Mandala Group

SUMMARY:
This study aims to investigate the effect of mandala coloring activity on test anxiety of nursing students.

DETAILED DESCRIPTION:
University life poses various challenges for students, such as being away from family, financial difficulties, and exam anxiety, which can increase stress levels. Test anxiety, a form of situation-specific anxiety, negatively impacts students' academic performance and well-being by reducing concentration and learning efficiency. The combination of theoretical and clinical demands in nursing education further amplifies stress, making it a particularly challenging field for students.

This study is a randomized controlled experimental research conducted between December 2, 2024, and January 13, 2025. The study population consists of nursing students enrolled in the Mental Health and Psychiatric Nursing course at a private university during the 2024-2025 academic year. Based on sample size calculations conducted using the G*Power program, considering similar studies and measurement methods, it was determined that 26 students per group are required. Accounting for potential data loss, it is planned to conduct the study with a total of 62 students, 32 in each group.

Students will be informed about the research, and those who voluntarily agree to participate will complete a "Demographic Characteristics Form" and a pre-test using the "Test Anxiety Inventory." Subsequently, students will be randomly assigned to the intervention and control groups in a 1:1 ratio using a random numbers table, with 31 students in each group. Students in the intervention group will be provided with mandala templates and coloring materials. They will be asked to color for 15 minutes twice a week over a two-month period. Email reminders will be sent to the students about the coloring sessions, and they will submit their completed mandalas to the researchers every Friday. Students who fail to complete two consecutive coloring sessions will be excluded from the study. Thirty minutes before the exam, the "Test Anxiety Inventory" will be applied as a post-test, and the study will be concluded. The data obtained will be subjected to statistical analysis, and the process of writing the manuscript will follow.

ELIGIBILITY:
Inclusion Criteria:

* Being a student enrolled in the Mental Health and Psychiatric Nursing course at the selected private university.
* Proficiency in the Turkish language.
* Having no physical disability that would hinder coloring activities.
* Willingness to participate voluntarily.

Exclusion Criteria:

* Students with psychological diagnoses such as anxiety or depression.
* Students who do not fully complete the questionnaire/survey forms.
* Students who neglect mandala coloring for two consecutive sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from test anxiety values at two hours | At the beginning of the study irst admission. Two months later.
  The items of the scale was created by including 50 anxiety statements developed by Baltaş (1999) with permission. The reliability analysis of the scale was conducted with the participation of 206 undergraduate students studying in Nursing, Physical Education Teaching, and Science Education departments. Data obtained from the application were subjected to factor analysis. As a result of the analysis, 12 items were removed from the scale due to factor load values being below 0.40, and 4 items were excluded for being non-discriminative (overlapping). The remaining 34 items were distributed across five sub-dimensions, with factor loadings ranging from 0.41 to 0.74. The scale is in a 5-point Likert format, and the internal reliability coefficient of the scale was calculated as Cronbach's Alpha (α) = 0.87.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze ACAVUT, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Sari Ozturk C, Kilicarslan Toruner E. The effect of mindfulness-based mandala activity on anxiety and spiritual well-being levels of senior nursing students: A randomized controlled study. Perspect Psychiatr Care. 2022 Oct;58(4):2897-2909. doi: 10.1111/ppc.13138. Epub 2022 Jul 3. PMID 35780483
- [Background] Khademi F, Rassouli M, Rafiei F, Moayedi S, Torres M, Marzban N, Haji E, Golitaleb M. The effect of mandala colouring on anxiety in hospitalized COVID-19 patients: A randomized controlled clinical trial. Int J Ment Health Nurs. 2021 Oct;30 Suppl 1(Suppl 1):1437-1444. doi: 10.1111/inm.12901. Epub 2021 Jun 18. PMID 34143568
- [Background] Zhang MQ, Liu X, Huang Y. Does Mandala Art Improve Psychological Well-Being in Patients? A Systematic Review. J Integr Complement Med. 2024 Jan;30(1):25-36. doi: 10.1089/jicm.2022.0780. Epub 2023 Sep 1. PMID 37668598